CLINICAL TRIAL: NCT03981250
Title: The ONE Study: Effect of One Minute of Resistance Exercise Per Day on Muscular Strength
Brief Title: Effect of One Minute of Resistance Exercise Per Day on Muscular Strength (The ONE Study)
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Professor Jason Gill, Professor, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 200180137
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Exercise
Keywords: Resistance training; Strength Training; Muscle Strength; voluntary failure
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial.
Masking Description: There is no masking due to intervention characteristics (exercise training programme).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group will be asked to keep their lifestyle behaviour and not increase their physical activity levels during the study period.
- Exercise Group (Experimental): The exercise group will engage in a home-based resistance exercise intervention for 12 weeks. They will perform 6 exercises, one each day for one minute, for 6 days a week.
  Interventions: Behavioral: 12-week home-based resistance exercise programme

INTERVENTIONS:
Behavioral: 12-week home-based resistance exercise programme — Participants will perform 6 exercises (press-ups, squats, squat jumps, plank, upright row and seated row) for one minute, aiming for the maximum number of repetitions. Participants will perform one exercise per day, for 6 days a week, for 12 weeks.
  Arms: Exercise Group

SUMMARY:
This study will evaluate the effect of one minute of resistance exercise per day on muscular strength in adults. Half of the participants will undergo a 12-week home-based resistance exercise programme, while the other half will continue their usual lifestyle behaviour.

DETAILED DESCRIPTION:
A resistance training programme can lead to a variety of health benefits including increases in muscle size and strength. Other potential health benefits of resistance training include reduction of body fat, increased metabolic rate, improve insulin sensitivity, blood glucose tolerance and blood lipid profiles. Meta-analyses indicate that while performing resistance exercise two or more times per week of resistance exercise per muscle group appears to be optimal to maximise strength gains, a single set of resistance exercise per muscle group per week, if performed to failure is sufficient to induce substantial strength changes.

The current physical activity guidelines recommend undertaking muscle strengthening activities involving major muscle groups two days a week or more, as well as undertaking at least 150 minutes per week of moderate intensity physical activity (or 75 minutes per week of vigorous intensity physical activity). However, only small portion of the population achieves the muscle strengthening aspect of the guidelines. As lack of time is often cited as a reason not to engage in physical activity, this study is seeking to investigate a low time-commitment approach to resistance exercise which could increase muscular strength. To address this, the present study will to split a typical single session of resistance exercise involving several exercises across different muscle groups into separate 1-minute micro-sessions where a different muscle group is exercised on each day of the week. The aim is to determine the effects of a one-minute-per-day home-based resistance exercise training on muscular strength.

The study is a randomized control trial in which the control group will continue their lifestyle behaviour and will be asked not to increase their physical activity levels and the exercise group will perform a 12-week home-based resistance exercise programme, involving doing one minute of resistance exercise per day on six days of the week, with a different exercise performed on each day. All participants will be measured at baseline, 4 weeks, 8 weeks and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years

Exclusion Criteria:

* Diabetes
* Uncontrolled hypertension (blood pressure > 150/90 on medication).
* History of cardiovascular disease
* Undertaking more than 150 minutes of moderate intensity or 75 minutes of vigorous physical activity or undertaking any resistance exercise.
* Other significant illness that would prevent the participant to undertake physical activity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2021-10-28 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle strength | Change between baseline and 4 weeks
  Change in 1-RM (one repetition maximum) (kg) for bench press, leg press and lat pull down (kg).
Muscle strength | Change between baseline and 8 weeks
  Change in 1-RM (one repetition maximum) (kg) for bench press, leg press and lat pull down (kg).
Muscle strength | Change between baseline and 12 weeks
  Change in 1-RM (one repetition maximum) (kg) for bench press, leg press and lat pull down (kg).

SECONDARY OUTCOMES:
Muscle endurance | Change between baseline and 4 weeks
  Change in maximal number of repetitions with a load of 50% of baseline 1-RM for bench press, leg press and lateral pull down.
Muscle endurance | Change between baseline and 8 weeks
  Change in maximal number of repetitions with a load of 50% of baseline 1-RM for bench press, leg press and lateral pull down.
Muscle endurance | Change between baseline and 12 weeks
  Change in maximal number of repetitions with a load of 50% of baseline 1-RM for bench press, leg press and lateral pull down.
Weight | Change between baseline and 4 weeks
  Change in weight (kg).
Weight | Change between baseline and 8 weeks
  Change in weight (kg).
Weight | Change between baseline and 12 weeks
  Change in weight (kg).
Waist | Change between baseline and 4 weeks
  Change in waist circumference (cm).
Waist | Change between baseline and 8 weeks
  Change in waist circumference (cm).
Waist | Change between baseline and 12 weeks
  Change in waist circumference (cm).
Body composition | Change between baseline and 4 weeks
  Change in fat mass and free fat mass measured by Bioelectrical Impedance Analysis (BIA).
Body composition | Change between baseline and 8 weeks
  Change in fat mass and free fat mass measured by Bioelectrical Impedance Analysis (BIA).
Body composition | Change between baseline and 12 weeks
  Change in fat mass and free fat mass measured by Bioelectrical Impedance Analysis (BIA).
Muscle thickness | Change between baseline and 12 weeks
  Change in muscle thickness of vastus lateralis (mm) measured with ultrasound.
Grip strength | Change between baseline and 4 weeks
  Change in grip strength (kg) measured using a hand grip dynamometer
Grip strength | Change between baseline and 8 weeks
  Change in grip strength (kg) measured using a hand grip dynamometer
Grip strength | Change between baseline and 12 weeks
  Change in grip strength (kg) measured using a hand grip dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Jason Gill, PhD, Principal Investigator — University of Glasgow
Locations (1):
- University of Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No